CLINICAL TRIAL: NCT02860650
Title: A Phase 1, First-in-human Study to Evaluate Safety, Tolerability, and Immunogenicity of Heterologous Prime-boost Regimens Using the Multivalent Filovirus Vaccines Ad26.Filo and MVA-BN-Filo Administered in Different Sequences and Schedules in Healthy Adult
Brief Title: A Study to Evaluate Safety, Tolerability, and Immunogenicity of Heterologous Prime-boost Regimens Using the Multivalent Filovirus Vaccines Ad26.Filo and MVA-BN-Filo Administered in Different Sequences and Schedules in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR108144; VAC69120FLV1001 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: AD26.Filo/MVA-BN-Filo or Placebo (Experimental): Participants will receive Ad26.Filo or placebo on Day 1 followed by MVA-BN-Filo or placebo on Day 57.
  Interventions: Biological: Ad26.Filo; Biological: MVA-BN-Filo; Biological: Placebo
- Group 2: MVA-BN-Filo/AD26.Filo or Placebo (Experimental): Participants will receive MVA-BN-Filo or placebo on Day 1 followed by Ad26.Filo or placebo on Day 57.
  Interventions: Biological: Ad26.Filo; Biological: MVA-BN-Filo; Biological: Placebo
- Group 3: MVA-BN-Filo/AD26.Filo or Placebo (Experimental): Participants will receive MVA-BN-Filo or placebo on Day 1 followed by Ad26.Filo or placebo on Day 15.
  Interventions: Biological: Ad26.Filo; Biological: MVA-BN-Filo; Biological: Placebo
- Subset of Group 3: AD26.Filo or Placebo (Experimental): The first 8 participants in Group 3 who are willing to enroll in the subset for third vaccination, will receive a third vaccination at Day 92. Participants who previously received placebo will receive placebo a third time and participants who previously received MVA-BN-Filo/Ad26.Filo vaccination will receive Ad26.Filo as third vaccination. After enrollment of the 8 participants, the unblinded monitor and unblinded pharmacist will assess whether 7 participants who previously received MVA-BN-Filo/Ad26.Filo vaccination have been enrolled. If less than 7 participants of the active vaccine regimen have been enrolled, 2 additional participants will be enrolled. If at least 7 participants of the active vaccine regimen have been enrolled, no further will be enrolled. The aim is to enroll 7 or 8 participants who will receive Ad26.Filo as third vaccination.
  Interventions: Biological: Ad26.Filo; Biological: Placebo
- Group 4: Ad26.ZEBOV/MVA-BN-Filo or placebo (Experimental): Participants will receive Ad26.ZEBOV or placebo on Day 1 followed by MVA-BN-Filo or placebo on Day 57.
  Interventions: Biological: Ad26.ZEBOV; Biological: Placebo; Biological: MVA-BN-Filo

INTERVENTIONS:
Biological: Ad26.Filo — Ad26.Filo intramuscular (IM) injection at a dose of 9*10^10 viral particles (vp).
  Arms: Group 1: AD26.Filo/MVA-BN-Filo or Placebo; Group 2: MVA-BN-Filo/AD26.Filo or Placebo; Group 3: MVA-BN-Filo/AD26.Filo or Placebo; Subset of Group 3: AD26.Filo or Placebo
Biological: MVA-BN-Filo — MVA-BN-Filo intramuscular (IM) injection at a dose of 5*10^8 infectious units (Inf U).
  Arms: Group 1: AD26.Filo/MVA-BN-Filo or Placebo; Group 2: MVA-BN-Filo/AD26.Filo or Placebo; Group 3: MVA-BN-Filo/AD26.Filo or Placebo
Biological: Ad26.ZEBOV — Ad26.ZEBOV intramuscular (IM) injection at a dose of 5*10^10 vp.
  Arms: Group 4: Ad26.ZEBOV/MVA-BN-Filo or placebo
Biological: Placebo — IM injection of 0.9 percent saline.
Biological: MVA-BN-Filo — MVA-BN-Filo intramuscular (IM) injection at a dose of 1*10^8 Inf U.
  Arms: Group 4: Ad26.ZEBOV/MVA-BN-Filo or placebo

SUMMARY:
The purpose of this study is to test the safety and immunogenicity of MVA-BN-Filo and Ad26.Filo as heterologous prime-boost vaccine regimens in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of greater than or equal to (>=) 18.5 and less than (<) 35.0 kilogram per square meter (kg/m^2)
* Healthy on the basis of physical examination, medical history, and the investigator's clinical judgment
* All women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) pregnancy test at screening, have a negative urine beta-hCG pregnancy test immediately prior to each study vaccine administration
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction from the start of screening onwards until at least 3 months after the last vaccination
* Participant must be available and willing to participate for the duration of the study visits and follow-up

Exclusion Criteria:

* Has been vaccinated with a candidate filovirus vaccine
* Has received any Ad26- or MVA-based candidate vaccines in the past
* Has been diagnosed with disease caused by Ebola virus (EBOV), Marburg virus (MARV), Sudan virus (SUDV), or Taï Forest virus (TAFV) or exposed to EBOV, MARV, SUDV, or TAFV, including participants who traveled to epidemic filovirus areas in West Africa during the last 2 years (that is, since the start of the last Ebolavirus outbreak) should be excluded from the study
* Chronic active hepatitis B or hepatitis C infection, documented by hepatitis B surface antigen and hepatitis C antibody, respectively
* Acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or body temperature greater than or equal to (>=) 38.0 degree Celsius on Day 1

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse events (AEs) | Up to 28 days after the last vaccination
Number of Participants With Reactogenicity (ie, Solicited Local and Systemic Adverse Events) | One Week after each study vaccine administration
Number of Participants With Serious Adverse Events | Up to the end of long-term follow-up (Day 360)

SECONDARY OUTCOMES:
Binding Antibody Responses Against Ebola Virus (EBOV), Marburg Virus (MARV), and Sudan Virus (SUDV) Glycoproteins (GPs) | Up to Day 360

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (1):
- Rockville, Maryland, United States

REFERENCES:
- [Derived] Bockstal V, Shukarev G, McLean C, Goldstein N, Bart S, Gaddah A, Anumenden D, Stoop JN, Marit de Groot A, Pau MG, Hendriks J, De Rosa SC, Cohen KW, McElrath MJ, Callendret B, Luhn K, Douoguih M, Robinson C. First-in-human study to evaluate safety, tolerability, and immunogenicity of heterologous regimens using the multivalent filovirus vaccines Ad26.Filo and MVA-BN-Filo administered in different sequences and schedules: A randomized, controlled study. PLoS One. 2022 Oct 5;17(10):e0274906. doi: 10.1371/journal.pone.0274906. eCollection 2022. PMID 36197845